CLINICAL TRIAL: NCT01749943
Title: Validation of a Hand-Held Dynamometer for Assessment of Lower Limb Muscle Strength in Multiple Sclerosis: Protocol for Strength Testing and Reliability Characteristics
Brief Title: Validation of Hand Held Dynamometer for Assessment of Lower Limb Muscle Strength in Multiple Sclerosis
Acronym: HHD
Status: Completed | Type: Observational
Sponsor: Brown, Theodore R., M.D., MPH (Individual)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: US-AVX-11-10213
Record Dates: First submitted 2012-11-26; First posted 2012-12-17 (Estimated); Last update posted 2013-08-22 (Estimated); Status verified 2013-08

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- EDSS Score 0-3.5: 21 Subjects Total : 7 with normal to mildly limited walking
- EDSS Score 4.0-5.5: 21 Subjects total: 7 subjects with moderately limited walking ability.
- EDSS Score 6.0-7.5: 21 Subjects total: 7 subjects with severely limited walking ability

SUMMARY:
Evaluate a method of testing the strength of five key lower limb muscle groups using a hand-held strength gauge (dynamometer).

DETAILED DESCRIPTION:
Purpose of this study is to assess the intra-rater and inter-rater reliability of a hand-held dynamometer (HHD) in the assessment of lower limb strength in patients with Multiple Sclerosis.

Also to establish a standardized strength testing procedure for key lower limb muscle groups using a HHD fo research and clinical purposes in Multiple Sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Stable patients with clinically definite Multiple Sclerosis
* No Multiple Sclerosis exacerbation 30 days prior to screening
* No change in disease modifying therapy for 30 day prior to screening

Exclusion Criteria:

* Inflammatory myopathy
* Endocarditis, pericarditis o rother unstable heart disease
* Cardiac surgery or myocardial infarction in the last 3 months
* Decompensated congestive heart failure
* Severe aortic stenosis
* Severe pulmonary hypertension
* Pulmonary embolus or infarction in the last 6 months
* Uncontrolled hypertension by history or by screening or baseline diastolic blood pressure >170 or systolic blood pressure >105
* Concomitant neurodegenerative neurological disease such as Amyotrophic Lateral Sclerosis (ALS) Parkinsons or hemiplegic stroke
* females who are pregnant
* Cognitive deficits that would interfere with the subjects's ability to give informed consent or preform study testing
* Painful orthopedic condition affecting the lower limbs
* Any other serious and/or unstable medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stable patients with clinically definite Multiple Sclerosis, aged 18 over, no Multiple Sclerosis exacerbation or change in disease modifying therapy for 30 days prior to screening. Subjects will fall into 1 of 3 EDSS catagories: 0-3.5; 4.0-5.5; 6.0-7.5.
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2012-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Assessment of HHD | Outcome measures will be assessed once we have captured all data points for all 21 subjects.
  To assess the intra-rater and inter-rater reliability of a hand-held dynamometer(HHD) in the assessment of lower limb strength in patients with Multiple Sclerosis.
  To establish a standardized strength testing procedure for key lower limb muscle groups using a HHD for research and clinical purposes in Multiple Sclerosis.

SECONDARY OUTCOMES:
Validation of a Hand-held dynamometer for assessment of lower limb muscle strength. | outcome measures will be assessed once we have captured all data points for all 21 subjects
  to establish a standardized strength testing procedure for key lower limb muscle groups using a Hand-held dynamometer for research and clinical purposes in Multiple Sclerosis.

CONTACTS AND LOCATIONS:
Overall Officials: Theodore R Brown, MD, Principal Investigator — MS Center at Evergreen Hospital
Locations (1):
- MS Center at Evergreen Hospital, Kirkland, Washington, United States